CLINICAL TRIAL: NCT07336264
Title: Characterization of Acute Nociceptive Pain and Analgesic Response in Pediatric and Adolescent Patients
Brief Title: Characterization of Acute Pain
Status: Recruiting | Type: Observational
Sponsor: Children's National Research Institute (Other)
Collaborators: VentureWell (Industry)
Responsible Party: Principal Investigator, Julia Finkel, Vice chief for Pain Medicine and Research, Children's National Research Institute
Other Study IDs: STUDY00001386; STUDY00001386 (Other: Childrens National IRB Protocol Number)
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Acute Pain, Postoperative; Postoperative Pain; Acute Pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Surgical Cohort: Children and adolescents ages 6 to 21 years undergoing elective surgical procedures (e.g., orthopedic or thoracic surgery) with no history of chronic pain prior to surgery. Participants will undergo non-invasive nociceptive measurements using the AlgometRx Nociometer at baseline and during postoperative follow-up, alongside standard clinical pain assessments. All pain management will follow standard of care and will not be influenced by study participation.
  Interventions: Device: AlgometRx Nociometer
- Bone Marrow Transplant (BMT) Cohort: Children and adolescents aged 6 to 21 years undergoing elective surgical procedures (e.g., orthopedic or thoracic surgery) with no history of chronic pain before surgery. Participants will undergo non-invasive nociceptive measurements using the AlgometRx Nociometer at baseline and during postoperative follow-up, alongside standard clinical pain assessments. All pain management will follow the standard of care and will not be influenced by study participation.
  Interventions: Device: AlgometRx Nociometer

INTERVENTIONS:
Device: AlgometRx Nociometer — The AlgometRx Nociometer is a non-invasive device used to measure nociceptive responses through neuroselective electrical stimulation and pupillometry. The device delivers low-intensity, painless electrical stimuli at specific frequencies to selectively activate sensory nerve fibers, while measuring stimulus-induced changes in pupil diameter. Data generated by the device are used or research measurement purposes only and do not guide or alter clinical care, treatment decisions,

SUMMARY:
This study aims to better understand how acute pain and responses to pain treatment can be measured in children and adolescents using a non-invasive device. Pain is usually assessed using self-reported or observational scales, which can be difficult to interpret, especially in pediatric patients. This study will evaluate whether a novel device, the AlgometRx Nociometer, can provide an objective measure of nociceptive pain. Participants ages 6 to 21 years who are undergoing elective surgery or bone marrow transplantation will be enrolled at Children's National Hospital. The device measures changes in pupil size in response to gentle electrical stimulation, which reflects activity in pain-related nerve pathways. Measurements will be taken before and after procedures and during routine hospital care, alongside standard pain assessments. This is an observational study. Participation will not change or guide any medical treatment, and all pain management will follow standard clinical care. The information collected may help improve future pain assessment and treatment for pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents ages 6 to 21 years
* Undergoing elective surgical procedures without a history of chronic pain, OR undergoing or planning to undergo bone marrow transplantation (BMT)
* Able to provide written informed assent and parental permission/consent, as applicable

Exclusion Criteria:

* Documented history of eye disease that precludes pupillometry
* Unwilling or unable to participate

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population includes children and adolescents ages 6 to 21 years receiving care at Children's National Hospital who are either undergoing elective surgical procedures or bone marrow transplantation. Participants will be followed prospectively and undergo non-invasive nociceptive measurements during routine clinical care, including periods before and after procedures and during inpatient follow-up. The study does not alter clinical management, and all treatments are provided according to standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-12-02 (Estimated); Study Completion 2028-06-02 (Estimated)

PRIMARY OUTCOMES:
Nociceptive Index | Baseline through up to 9 weeks of follow-up
  The nociceptive index calculated from neuroselective stimulus-induced pupillary reflex dilation (nPRD) measurements obtained using the AlgometRx Nociometer. The index is derived from the area under the curve (AUC) of pupillary dilation responses corresponding to selective activation of sensory nerve fiber types and is used to characterize acute nociceptive pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in publications, including nociceptive index measurements, standard pain assessment scores, and relevant clinical variables. Direct identifiers will not be shared.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Instrument: PROMIS Pain Intensity - Short Form 3a v1.0 | NIDA CTN Common Data Elements. https://cde.nida.nih.gov/instrument/0a481bfb-a5e6-3c84-e050-bb89ad43314d
- [Background] Page MG, Katz J, Stinson J, Isaac L, Martin-Pichora AL, Campbell F. Validation of the numerical rating scale for pain intensity and unpleasantness in pediatric acute postoperative pain: sensitivity to change over time. J Pain. 2012 Apr;13(4):359-69. doi: 10.1016/j.jpain.2011.12.010. Epub 2012 Mar 15. PMID 22424915
- [Background] Wong-Baker FACES® Pain Rating Scale. (2016)
- [Background] Lavoie Smith EM, Li L, Hutchinson RJ, Ho R, Burnette WB, Wells E, Bridges C, Renbarger J. Measuring vincristine-induced peripheral neuropathy in children with acute lymphoblastic leukemia. Cancer Nurs. 2013 Sep-Oct;36(5):E49-60. doi: 10.1097/NCC.0b013e318299ad23. PMID 23842524
- [Background] Barr MS, Farzan F, Davis KD, Fitzgerald PB, Daskalakis ZJ. Measuring GABAergic inhibitory activity with TMS-EEG and its potential clinical application for chronic pain. J Neuroimmune Pharmacol. 2013 Jun;8(3):535-46. doi: 10.1007/s11481-012-9383-y. Epub 2012 Jun 29. PMID 22744222
- [Background] Chouchou F, Perchet C, Garcia-Larrea L. EEG changes reflecting pain: is alpha suppression better than gamma enhancement? Neurophysiol Clin. 2021 Jun;51(3):209-218. doi: 10.1016/j.neucli.2021.03.001. Epub 2021 Mar 16. PMID 33741256
- [Background] Crawford L, Mills E, Meylakh N, Macey PM, Macefield VG, Henderson LA. Brain activity changes associated with pain perception variability. Cereb Cortex. 2023 Mar 21;33(7):4145-4155. doi: 10.1093/cercor/bhac332. PMID 36069972
- [Background] Minetama M, Kawakami M, Teraguchi M, Matsuo S, Enyo Y, Nakagawa M, Yamamoto Y, Nakatani T, Sakon N, Nagata W, Nakagawa Y. MRI grading of spinal stenosis is not associated with the severity of low back pain in patients with lumbar spinal stenosis. BMC Musculoskelet Disord. 2022 Sep 12;23(1):857. doi: 10.1186/s12891-022-05810-y. PMID 36096768
- [Background] Fomberstein K, Qadri S, Ramani R. Functional MRI and pain. Curr Opin Anaesthesiol. 2013 Oct;26(5):588-93. doi: 10.1097/01.aco.0000433060.59939.fe. PMID 23995063